CLINICAL TRIAL: NCT02807051
Title: A Phase 1, Open-Label, Drug-Interaction Study to Evaluate the Effect of Clarithromycin, a Potent CYP3A4 Inhibitor, on the Systemic Exposure of Pacritinib in Healthy Subjects
Brief Title: To Evaluate the Effect of Clarithromycin on the Systemic Exposure of Pacritinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PAC104
Record Dates: First submitted 2016-05-03; First posted 2016-06-21 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Drug Interaction Study
MeSH Terms: interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Clarithromycin

ARMS (1):
- Pacritinib and Clarithromycin (Experimental): Single 400-mg (four 100-mg capsules; lot number 21341) oral doses of pacritinib were administered in the fasted state on Days 1 and 12. Twice daily, 500-mg (1 tablet) oral doses of clarithromycin were administered with or without food on Days 8 through 11 and in the fasted state on the morning of Day 12
  Interventions: Drug: Pacritinib; Drug: Clarithromycin; Drug: Pacritinib and Clarithromycin

INTERVENTIONS:
Drug: Pacritinib — Single 400-mg dose (four 100-mg capsules) administered in the morning on Days 1 and 12
  Other Names: Pacritinib 100mg
Drug: Clarithromycin — Twice-daily, 500-mg dose (one 500-mg tablet) administered every 8 to 12 hours on Day 8 through the morning of Day 12
  Other Names: Clarithromycin 500mg
Drug: Pacritinib and Clarithromycin — On Day 12, a single oral 400-mg dose of pacritinib was co-administered with the final 500-mg dose of clarithromycin
  Other Names: Pacritinib 100mg and Clarithromycin 500mg

SUMMARY:
This will be an open-label, single-center, crossover, one-way, drug-interaction study to evaluate the effect of 500 mg clarithromycin BID (dosed to steady state) on the PK of a single 400-mg dose of pacritinib in healthy male and female subjects.

DETAILED DESCRIPTION:
This was a single-center, open-label, one-way crossover, drug-interaction study. On Day 1, subjects received a single oral 400-mg dose of pacritinib. On Day 8 through the morning of Day 12, following a 7-day washout period, 500-mg oral doses of clarithromycin were administered twice daily (BID), 8 to 12 hours apart. It was anticipated that steady-state concentrations of clarithromycin would be achieved by Day 12. On Day 12, a single oral 400-mg dose of pacritinib was co-administered with the final 500-mg dose of clarithromycin.

ELIGIBILITY:
Inclusion Criteria:

1. males or females, between 18 and 55 years of age, inclusive;
2. BMI between 18.5 and 32.0 kg/m2, inclusive;
3. in good health, determined by no clinically significant findings from medical history, physical examination, and vital signs;
4. clinical laboratory evaluations (including clinical chemistry panel [fasted at least 10 hours], CBC, and UA) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator;
5. negative test for selected drugs of abuse (including alcohol) at Screening and at Check-in;
6. negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV]) and negative HIV antibody screens;
7. females of childbearing potential must be non-pregnant and non-lactating, and agree to use contraception from the time of signing the informed consent or 10 days prior to Check-in (Day -1) until 30 days after the final dose administration. One of the following forms of contraception must be used from the time of signing the informed consent or 10 days prior to Check-in (Day -1) until 30 days after the final dose administration: non-hormonal intrauterine device (IUD) with spermicide; female condom with spermicide; contraceptive sponge with spermicide; intravaginal system (eg, NuvaRing®); diaphragm with spermicide; cervical cap with spermicide; male sexual partner who agrees to use a male condom with spermicide; sterile sexual partner; or abstinence. Oral, implantable, transdermal, or injectable hormonal contraceptives may not be used from the time of signing the informed consent or 10 days prior to Check-in (Day -1) until 14 days after the final dose administration. For all females, the pregnancy test result must be negative at Screening and Check-in (Day -1). Females not of childbearing potential must be postmenopausal for at least 1 year or surgically sterile (eg, tubal ligation, hysterectomy) for at least 90 days;
8. males will either be surgically sterile (ie, vasectomy, documented in the medical record by a physician) or agree to use from Check-in (Day -1) until 90 days following Study Completion (Day 19)/ET, one of the following approved methods of contraception: male condom with spermicide; sterile sexual partner; or use by female sexual partner of an IUD with spermicide, a female condom with spermicide, a contraceptive sponge with spermicide, an intravaginal system, a diaphragm with spermicide, a cervical cap with spermicide, or oral, implantable, transdermal, or injectable contraceptives. Subjects must agree to refrain from sperm donation from Check-in (Day -1) until 90 days following Study Completion (Day 19)/ET;
9. able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. history or clinical manifestation of clinically significant cardiovascular, pulmonary, hepatic (eg, hepatitis), renal, hematologic, gastrointestinal (eg, celiac disease, peptic ulcer, gastroesophageal reflux, inflammatory bowel disease), metabolic, allergic, dermatological, neurological, or psychiatric disorder (as determined by the Investigator; appendectomy and cholecystectomy are not considered to be clinically significant disease);
2. abnormalities in liver function tests (any/all of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase >1.5 × upper limit of normal [ULN]; gamma-glutamyl transferase >2 × ULN; or total bilirubin >1.3 × ULN) or kidney function tests (serum creatinine > ULN) that are considered clinically significant by the Investigator, in consultation with the Sponsor;
3. history of malignancy, except the following; cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps;
4. history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, including clarithromycin, unless approved by the Investigator;
5. history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and hernia repair will be allowed;
6. history of Gilbert's Syndrome;
7. history or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant; QTcF >450 msec, or factors that increase risk for QTc interval prolongation (eg, heart failure, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], or family history of long QT interval syndrome)
8. history of alcoholism or drug addiction within 1 year prior to Check-in (Day -1);
9. use of tobacco- or nicotine-containing products within 6 months prior to Check-in (Day -1) and during the entire study;
10. consumption of alcohol- or caffeine-containing foods and beverages for 72 hours prior to Screening and during the entire study;
11. consumption of grapefruit-containing foods and beverages or other CYP3A4 inhibitors or inducers for 72 hours prior to Screening and during the entire study
12. participation in any other investigational drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days prior to Check-in (Day -1), whichever is longer;
13. use of oral, implantable, injectable, or transdermal hormonal contraceptives within 10 days prior to Check-in (Day -1) or from the time of signing the informed consent (females only) until 14 days after the final dose administration;
14. use of any prescription medications and/or products within 14 days prior to Check-in (Day -1) and during the entire study, unless deemed acceptable by the Investigator in consultation with the Sponsor;
15. use of any over-the-counter, non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in (Day -1) and during the entire study, unless deemed acceptable by the Investigator;
16. poor peripheral venous access;
17. donation of blood from 30 days prior to Screening through Study Completion (Day 19)/ET, inclusive, or of plasma from 2 weeks prior to Screening through Study Completion (Day 19)/ET, inclusive;
18. receipt of blood products within 2 months prior to Check-in (Day -1);
19. any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Estimate ratios of geometric mean values and the corresponding 90% confidence intervals (CIs) for pacritinib treatments with and without clarithromycin | Fifteen days approximately
  To estimate ratios of geometric mean values and the corresponding 90% confidence intervals

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | from Day 1 to Day 19
  To evaluate the safety of pacritinib and tolerability of a single 400 mg dose of pacritinib in patients with hepatic impairment. Safety endpoints for this study include AEs, vital signs, clinical laboratory evaluations, physical examinations, and single 12-lead ECGs
The apparent terminal elimination rate constant (λZ) and the respective apparent terminal elimination half-life (t½). | Plasma (Day 1 and 12): 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
The maximum plasma concentration (Cmax). | Plasma (Day 1 and 12): 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To characterize the pharmacokinetic (PK) profile of pacritinib and its major human metabolites following single-dose administration with and without concomitant clarithromycin in healthy subjects
The time to reach maximum plasma concentration (tmax). | Plasma (Day 1 and 12): 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To characterize the pharmacokinetic (PK) profile of pacritinib and its major human metabolites following single-dose administration with and without concomitant clarithromycin in healthy subjects
The area under the plasma concentration-time curve from time zero to time of the last measured concentration above the limit of quantification (AUC0-t) | Plasma (Day 1 and 12): 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  To characterize the pharmacokinetic (PK) profile of pacritinib and its major human metabolites following single-dose administration with and without concomitant clarithromycin in healthy subjects
The area under the plasma concentration-time curve from zero to infinity (AUC0-∞). | Plasma (Day 1 and 12): 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
The apparent volume of distribution (Vd). | Plasma (Day 1 and 12): 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
The apparent total body clearance (CL/F). | Plasma (Day 1 and 12): 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Frank Farmer, MD, PhD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes